CLINICAL TRIAL: NCT06209749
Title: Pembangunan Dan Keberkesanan Modul Intervensi Berasaskan Sensori Dalam Kalangan Kanak-kanak Dengan Autisme / The Development and Effectiveness of Sensory-based Intervention Modules in Children With Autism Spectrum Disorders
Brief Title: Keberkesanan Modul Intervensi Berasaskan Sensori Dalam Kalangan Kanak-kanak Dengan Autisme/The Effectiveness of Sensory-based Intervention in Children With Autism Spectrum Disorders.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Ministry of Education, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JEP-2022-576
Record Dates: First submitted 2023-12-07; First posted 2024-01-17 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Sensory-based intervention; Social skills; Play; Children
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Sensory-based intervention module will be given for three sessions a week for 12 weeks (30 minutes per session).
  Usual school activities will be given four days a week for 12 weeks (6 hours per day)
  Interventions: Other: Sensory-based intervention module
- Control group (No Intervention): Usual school activities will be given four days a week for 12 weeks (6 hours per day)

INTERVENTIONS:
Other: Sensory-based intervention module — Consists of sensory-based activities (Set A-F) with six weeks of individual sessions and six weeks of group sessions
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of Sensory-based intervention modules on children with Autism Spectrum Disorder (ASD). The main questions this study aims to answer is How do children with ASD respond to Sensory-based intervention (SBI) in terms of their sensory processing, social skills, and play? Thus, the objective of this study is to determine the significant differences in sensory processing, social skills, and play in children with ASD before and after receiving the Sensory-based intervention (SBI) module in the intervention and control groups.

Participants in this study are children with ASD, aged between 4-6 years, who attend Pusat PERMATA Kurnia, a specialized school for ASD. The children will undergo assessments using the Sensory Profile 2 and Sensory Processing Measurement 2 for sensory processing, the Social Responsiveness Scale for social skills, and Knox Preschool Play Scale to measure play.

Researchers will compare two groups: one receiving Sensory-Based Interventions (SBI) modules with usual school activities (intervention group), and the other receiving only usual school activities (control group). We aim to see if the SBI module makes a significant difference in sensory processing, social skills, and play in children with ASD.

DETAILED DESCRIPTION:
The proposed research design for this study is a quantitative approach using a Randomized Controlled Trial (RCT) method. This design randomly assigns participants to either an experimental or a control group, utilizing an application for allocation. The study includes pre-tests, post-tests and follow-ups to measure dependent variables such as sensory processing, social skills, and play.

For sampling, the study will be conducted at Pusat PERMATA Kurnia, a school and research centre specialized for children with Autism Spectrum Disorder (ASD). The participants will be children with ASD, aged 4-6 years, attending learning sessions at Pusat PERMATA Kurnia. The sampling method used is simple random sampling using the Research Randomizer application on the internet. This double-blind study involves occupational therapists who meet the criteria and will be informed about the study without knowing the group allocation.

The sample size is calculated based on phase 3 study objectives using G power software, considering an alpha level of 0.05 and a power of 0.8. As per the calculations, the total sample size for this effectiveness study is 32 participants, accounting for the largest dependent variable size in both intervention and control groups.

The inclusion criteria for the sample are children with ASD:

i. whose diagnosis of ASD is confirmed by a Medical Officer) ii. aged 4-6 years, and iii. experiencing sensory processing disorders (seeking, hypersensitive and under responsiveness) as screened using Sensory Profile 2.

The exclusion criteria for the sample are children with ASD:

i. Attend any other occupational therapy intervention at Pusat PERMATA Kurnia or outside ii. Have chronic medical problems such as heart problems or asthma

Data collection involves screening and procedure steps. Researchers will screen for potential participants based on inclusion and exclusion criteria. Two occupational therapists who are Malaysian citizens and have experience managing children with ASD will be appointed for the intervention. One occupational therapist who was not doing intervention was assigned as an assessor in assessments which is double-blind to the study groups. The intervention group will receive a Sensory-based intervention module and usual school activities thrice a week for 12 weeks duration. The control group will receive school activities learning four times a week for 12 weeks without the SBI module. Post-tests will be conducted after the intervention period and follow-up test after 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Occupational Therapist

   a. Implements SBI intervention
2. Children with ASD

   1. A Medical Officer confirms the diagnosis of ASD
   2. Aged 4-6 years
   3. Experiencing a sensory processing disorder
   4. Get the usual school activities

Exclusion Criteria:

1. Occupational Therapist

   a. Non-citizen
2. Children with ASD

   1. Attend any other occupational therapy intervention at Pusat PERMATA Kurnia or outside
   2. Have chronic medical problems such as heart problems or asthma

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
32 participants will assess sensory processing using Sensory Profile 2 | 1st week (Pre-test), 14th week (Post-test) and 18th week (Follow up)
  The Sensory Profile™ 2 family of assessments provides standardized tools to help evaluate a child's sensory processing patterns in the context of home, school, and community-based activities. Parents or caregivers are assessing this form. This form can be used from newborn until 14:11 years. This form consists of 86 Likert-type items rated in terms of the frequency of a specific behaviour (0=Does do not apply, 1=Almost never, 2=Occasionally, 3=Half of the time, 4=Frequently, 5=Almost always) and require about 15-20 minutes to complete. Test-retest :0.83-0.97, Inter-rater: 0.70-0.90, Internal consistency 0.57-0.93
32 participants will assess sensory processing using Sensory Processing Measurement 2 (SPM-2) | 1st week (Pre-test), 14th week (Post-test) and 18th week (Follow up)
  SPM-2 forms are designed to assess sensory functioning, praxis, and social participation across the lifespan, with unique forms in each of the five age levels. In this study, we used Child SPM-2 (5-12 years). This form consists of a Home form (Completed by parents or another caregiver) and a School Form (completed by the child's primary classroom teacher or aide). This form consists of 80 Likert-type items rated regarding the frequency of a specific behaviour (1=Never,2= Occasionally, 3=Frequently, 4=Always). It requires about 20 to 30 minutes to complete-higher scores representing more problematic behavior. Evidence supporting reliability included median estimates of internal consistency of 0.86, test-retest reliability of 0.84, alternate-forms reliability of 0.78, and interrater reliability of 0.66.
32 participants will assess social skills using Social Responsiveness Scale 2 (SRS-2) | 1st week (Pre-test), 14th week (Post-test) and 18th week (Follow up)
  SRS-2 is a 65-item Likert scale with the objective measure of symptoms associated with autism-related components of social impairment. This form allows ratings to be collected on individuals across the age span from 2.5 years through adulthood. This study used the School Age (ages 4 to 18 years) rate by parents and teachers. Raters can complete the 65 items in 15-20 minutes. Scoring (1=not true, 2=sometimes true, 3=often true, 4=almost always true) with higher scores represents more social impairment in autistic children. Test-retest: 0.83-0.97, Inter-rater 0.72-0.91, Internal consistency 0.95
32 participants will assess play skills using Knox Preschool Play Scale | 1st week (Pre-test), 14th week (Post-test)
  Knox Preschool Play Scale is an observational assessment designed to give a developmental description of typical play behavior from birth through the age of 6 years. The items are grouped into four dimensions. Reviewing existing developmental and play scales determined the behavior descriptions under each dimension. The observation is in the range of 30-60 minutes. Within the factors, the observer places a mark above each descriptor each time it is observed. Then, the factor is ranked at the highest level unless the descriptor is insignificant. Scoring ( 0-6 months, 6-12 months, 12-18 months, 18-24 months, 24-30 months, 30-36 months, 36-48 months, 48-60 months, 60-72 months). Each factor is scored at the upper age of the age grouping. To achieve each dimension, the observer takes the mean of the factor scores. To cut an overall play age, the observer takes the mean of the dimension scores. Test-retest: 0.86-0.96, Inter-rater 0.89-0.98, Internal consistency 0.95.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusat PERMATA Kurnia, Sentul, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No